CLINICAL TRIAL: NCT06122363
Title: The Impact of Incomplete Endometrial Ablation on the Success Rate of Novasure Endometrial Ablation
Brief Title: Impact of Incomplete Endometrial Ablation
Status: Active, not recruiting | Type: Observational
Sponsor: Maxima Medical Center (Other)
Responsible Party: Principal Investigator, Danique Roelen, Medical student, Maxima Medical Center
Other Study IDs: Incomplete Novasure ablation
Record Dates: First submitted 2023-11-05; First posted 2023-11-08 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Heavy Menstrual Bleeding
MeSH Terms: conditions — Menorrhagia | interventions — Hysteroscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Complete Novasure endometrial ablation: After treatment with novasure, the hysteroscopy showed no remains of endometrium, , so a complete novasure endomentrial ablation
  Interventions: Device: hysteroscopy
- Incomplete Novasure endometrial ablation: After treatment with novasure, the hysteroscopy showed remains of endometrium, so an incomplete novasure endomentrial ablation
  Interventions: Device: hysteroscopy

INTERVENTIONS:
Device: hysteroscopy — uterine hysteroscopy right after Novasure endometrial ablation

SUMMARY:
The aim of the proposed protocol is to study the impact of incomplete endometrial ablation on the PBAC score, reintervention, satisfaction, controlled bleeding and dysmenorrhea at 24 months after Novasure endometrial ablation, in women with heavy menstrual bleeding treated at Máxima Medical Centre Veldhoven, in The Netherlands.

DETAILED DESCRIPTION:
The primary outcome is blood loss at 24 months after treatment, measured with the PBAC-score according to Higham. To calculate this score women were asked, in the MIRA and MIRA2 study, to record their menstrual blood loss for one month counting the number of super tampons or pads used each day. The total score was calculated using a score of 1 for each lightly saturated tampons. For pads the scores were respectively 1, 5 and 20. Secondary outcome measures were controlled bleeding, defined as a PBAC-score not exceeding 75 points, PBAC score of zero, re-intervention rate 24 months after treatment, satisfaction with treatment (measured with a 5-point Likert scale) and dysmenorrhea.

In addition, multiple variables were analyzed in predicting the occurrence of incomplete endometrial ablation, including age, BMI, cavum length, cavum width, ablation time, ablation power, nulliparity, sterilization in history, section caesarea in history, position of the uterus (AVF/RVF), presence of myomas, the presence of adenomyosis and surgery under local anesthesia, generally without sterilization or generally in combination with sterilization. Information was collected from EPD and the MIRA and MIRA2 databases.

ELIGIBILITY:
Inclusion Criteria:

* Endometrial ablation between 2012 and 2023 in Máxima Medical Centre
* Women had to suffer from heavy menstrual bleeding

Exclusion Criteria:

- No saved hysteroscopy images or bad quality hysteroscopy images

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — men can not suffer from heavy menstrual bleeding
Study Population: This retrospective cohort study was carried out using the data of women who participated in the MIRA study and the MIRA2 study including RCT and prospective cohort database. These women have given informed consent for their data to be used for future research into treatments for heavy menstrual bleeding. To be eligible for study inclusion, women had to suffer from heavy menstrual bleeding, and have undergone Novasure endometrial ablation at Máxima MC between January 2012 and July 2023. Women were excluded from the database if the hysteroscopy images were not saved, or these images were of poor quality.
Sampling Method: Non-Probability Sample
Enrollment: 121 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Pictorial Blood Assessment Chart (PBAC) score | 24 months
  Blood loss of 1 month, measured by the number of needed tampons/pads and how heavily they are filled with blood. The higher the score, the more severe blood loss. From 150 points the amount is defined as heavy menstrual bleeding.

SECONDARY OUTCOMES:
Rate of reintervention | 24 months
  Surgical and Medical reintervention
Dysmennorrhea | 24 months
  Presence of dysmennorrhea. Categorized as absence, mild, moderate and severe.
Number of patients having controlled bleeding | 24 months
  Pictorial Blood Assessment Chart (PBAC) score less than 75.
Satisfaction of the patient with the treatment | 24 months
  Satisfaction measured with a 5-point Likert scale. 1=very unsatisfied, 2= unsatisfied, 3= neutraal, 4= satisfied, 5= very satisfied.

OTHER OUTCOMES:
Number of possible prognostic variables predicting the occurrence of incomplete endometrial ablation. | baseline
  Age, BMI, cavum length, cavum width, ablation time, ablation power, nulliparity, sterilization in history, section caesarea in history, position of the uterus (AVF/RVF), presence of myomas, the presence of adenomyosis and surgery under local anesthesia, generally without sterilization or generally in combination with sterilization

CONTACTS AND LOCATIONS:
Overall Officials: Marlies M.Y. Bongers, PhD, MD, Principal Investigator — Maxima Medical Center
Locations (1):
- Máxima MC, Veldhoven, North Brabant, Netherlands